CLINICAL TRIAL: NCT02414906
Title: Goal Directed Therapy in the Early Phase of Acute Kidney Injury in Critical Ill Patients
Brief Title: Goal Directed Therapy for Acute Kidney Injury in Critical Ill Patients
Acronym: GDT-AKIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: Hospital de Base (Other); Hospital do Servidor Publico Estadual (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Prata Amendola, MD, Barretos Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BarretosCH-UTI 1
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Acute Kidney Injury
Keywords: Goal Directed Therapy; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Goal-directed therapy
  Interventions: Other: Goal-directed therapy
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Goal-directed therapy — Goal-directed therapy with fluids and dobutamine
  Other Names: Protocol of ressuscitation
  Arms: Intervention group

SUMMARY:
Acute kidney injury (AKI) is a frequent complication in critically ill patients admitted to intensive care unit (ICU) and it is associated with increased morbimortality.

There is evidence that perioperative hemodynamic optimization decreases the incidence of AKI in the post operative phase in high-risk patients. We aimed to evaluate if the use of a goal-directed therapy to increase oxygen delivery in the early phase of acute kidney injury can decrease the prevalence of patients with acute renal failure.

DETAILED DESCRIPTION:
Randomized, controlled, multicenter study.The intervention group was monitored with Flo Trac/Vigileo and optimized with fluid challenges, dobutamine and blood transfusion, if necessary, to maintain a IDO² ≥600ml/min/m² during 8h. The control group was treated according to the discretion of the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the Intensive Care Unit with Acute Kidney Injury (AKI) classified as AKIN 1 (increase in serum creatinine ≥0.3 mg/dL and/or urine output less than 0.5 ml/kg/h over 6 hours) for less than 12 hours.

Exclusion Criteria:

* ICU length of stay >10 days, nefrectomy, chronic kidney disease undergoing hemodialysis, baseline creatinine ≥4 mg/dL, life expectance ≤ than 1 month, pregnancy, severe arrhythmia, severe heart failure (≤ III, NYHA), acute myocardial infarction (AMI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
acute kidney injury | 2 months

SECONDARY OUTCOMES:
death | 2 months

OTHER OUTCOMES:
lenght of stay | 2 months

REFERENCES:
- [Derived] Amendola CP, Silva-Jr JM, Carvalho T, Sanches LC, Silva UVAE, Almeida R, Burdmann E, Lima E, Barbosa FF, Ferreira RS, Carmona MJC, Malbouisson LMS, Nogueira FAM, Auler-Junior JOC, Lobo SM. Goal-directed therapy in patients with early acute kidney injury: a multicenter randomized controlled trial. Clinics (Sao Paulo). 2018 Oct 29;73:e327. doi: 10.6061/clinics/2018/e327. PMID 30379222